CLINICAL TRIAL: NCT04623489
Title: ¡Vivir Mi Vida!: A Pilot Study of a Lifestyle Intervention to Optimize Health Outcomes in Latino Patients
Brief Title: ¡Vivir Mi Vida! Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Antelope Valley Partners for Health (Other); Wesley Health Centers - Antelope Valley (Unknown)
Responsible Party: Principal Investigator, Stacey Lynn Schepens Niemiec, Associate Professor of Research, University of Southern California
Masking: None
Other Study IDs: HS-14-00725
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Healthy Lifestyle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: ¡Vivir Mi Vida! Lifestyle Intervention
  Other Names: VMV

SUMMARY:
Rationale: By the year 2050, the number of older adults in the US will more than double. Because older adults are more likely to develop chronic conditions such as cardiovascular disease and arthritis, society is facing a healthcare crisis if effective ways to prevent such diseases is not found. This is especially urgent for Latinos because they are the nation's fastest growing ethnic group and they are in many cases at greater risk for chronic disease. Objectives: ln this proposed pilot project, the goal is to understand if a lifestyle intervention - iVivir Mi Vida! (iVMV!) - is feasible, acceptable, and shows preliminary promise in helping late middle-aged Latinos experience better health. The investigators will accomplish this goal by pilot testing the implementation of iVMV! in collaboration with community health service partners in Antelope Valley. Methods: ln this study, 40 patients, aged 50-65 years who are enrolled in Antelope Valley health centers will receive the iVMV! lifestyle-based health program. This program lasts four months and will be delivered by promotores (respected lay heath workers from the Latino community). Intervening promotores will be supervised by an occupational therapist and a senior promotora. Within the program, patients will participate in small group sessions at their local community healthcare facilities and will also receive numerous visits from the promotores in their homes. The program will involve weekly sessions in which the participants will be taught how to practice healthy lifestyle choices, such as exercising, eating healthy food, and reducing stress. Initially and at the end of the four-month program, the investigators will measure health outcomes such as self-rated quality of life, diet and exercise, cholesterol and glucose levels, blood pressure, and weight. The investigators will also ask participants, promotores, and other research staff about their overall experiences during the study so that the investigators can improve our program for the future. Mixed-methods procedures will be used to analyze qualitative data (e.g., interview transcripts) and quantitative data (e.g., pre-post intervention health outcomes and 12-month follow-up). Anticipated lmpact: The study will provide critical information about the feasibility and acceptability and preliminary data on the health impact of the iVMV! intervention on late middle-aged Latino adults who are at risk for disease. Information collected from this study will inform the design of a larger-scale implementation study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged at least 50 years at the outset of the four-month intervention and will be no older than 65 years upon completion of the intervention
2. Self-identify as Latino/Hispanic
3. Are fluent in Spanish
4. Live in Antelope Valley and do not plan on moving within six months from the beginning of the study
5. Are enrolled as a patient in the Antelope Valley Community Clinic
6. Have visited his/her primary care healthcare facility within the past year
7. Will be available by telephone for the duration of the intervention
8. Are oriented to person, place, and time as tested by asking the person's name, date, age, and place of residence
9. Self-report their ability to participate for the duration of the intervention

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2015-12-28 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 4 months on the Measure Yourself Medical Outcome Profile (MYMOP2) | 4 months
  Comprised of an overall profile score and four symptom/well-being subscales. Individuals identified one to two currently bothersome symptoms. They rated each symptom's severity and how much it interfered with daily activities. They also rated their overall well-being.
  MYMOP Profile Scores can be calculated as a mean of the ratings. These have values between 0 and 6; the higher the score, the worse the outcome. A decrease in scores is considered improvement.
Change from baseline to 16 months on the Measure Yourself Medical Outcome Profile (MYMOP2) | 16 months
  Comprised of an overall profile score and four symptom/well-being subscales. Individuals identified one to two currently bothersome symptoms. They rated each symptom's severity and how much it interfered with daily activities. They also rated their overall well-being.
  MYMOP Profile Scores can be calculated as a mean of the ratings. These have values between 0 and 6; the higher the score, the worse the outcome. A decrease in scores is considered improvement.
Change from 4 months to 16 months on the Measure Yourself Medical Outcome Profile (MYMOP2) | 16 months
  Comprised of an overall profile score and four symptom/well-being subscales. Individuals identified one to two currently bothersome symptoms. They rated each symptom's severity and how much it interfered with daily activities. They also rated their overall well-being.
  MYMOP Profile Scores can be calculated as a mean of the ratings. These have values between 0 and 6; the higher the score, the worse the outcome. A decrease in scores is considered improvement.

SECONDARY OUTCOMES:
Change from baseline to 4 months on the PROMIS Satisfaction with Participation in Social Roles - Short Form 7a | 4 months
  Satisfaction with performing usual social roles and activities
Change from baseline to 16 months on the PROMIS Satisfaction with Participation in Social Roles - Short Form 7a | 16 months
  Satisfaction with performing usual social roles and activities
Change from 4 months to 16 months on the PROMIS Satisfaction with Participation in Social Roles - Short Form 7a | 16 months
  Satisfaction with performing usual social roles and activities
Change from baseline to 4 months on the Pittsburgh sleep quality index (PSQI) | 4 months
  Global sleep quality, sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medications, and daytime dysfunction.
  The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points. In all cases, a score of 0 indicates no difficulty, whereas a score of 3 indicates severe difficulty. The seven component scores are then added to yield one global score, with a range of 0-21 points, 0 indicating no difficulty and 21 indicating severe difficulties in all areas.
Change from baseline to 16 months on the Pittsburgh sleep quality index (PSQI) | 16 months
  Global sleep quality, sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medications, and daytime dysfunction.
  The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points. In all cases, a score of 0 indicates no difficulty, whereas a score of 3 indicates severe difficulty. The seven component scores are then added to yield one global score, with a range of 0-21 points, 0 indicating no difficulty and 21 indicating severe difficulties in all areas.
Change from 4 months to 16 months on the Pittsburgh sleep quality index (PSQI) | 16 months
  Global sleep quality, sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medications, and daytime dysfunction.
  The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points. In all cases, a score of 0 indicates no difficulty, whereas a score of 3 indicates severe difficulty. The seven component scores are then added to yield one global score, with a range of 0-21 points, 0 indicating no difficulty and 21 indicating severe difficulties in all areas.
Change from baseline to 4 months on the Single item stress index | 4 months
  General level of stress 'these days' The response was recorded on a 5-point Likert scale varying from 1 "not at all" to 5 "very much." Higher score is worse stress.
Change from baseline to 16 months on the Single item stress index | 16 months
  General level of stress 'these days' The response was recorded on a 5-point Likert scale varying from 1 "not at all" to 5 "very much." Higher score is worse stress.
Change from 4 months to 16 months on the Single item stress index | 16 months
  General level of stress 'these days' The response was recorded on a 5-point Likert scale varying from 1 "not at all" to 5 "very much." Higher score is worse stress.
Change from baseline to 4 months on the International Physical Activity Questionnaires (IPAQ) | 4 months
  Vigorous activity, moderate activity, walking, and time spent sitting.
  There are two forms of output from scoring the IPAQ. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity. Higher activity levels or more MET minutes per week equates to more physical activity.
Change from baseline to 16 months on the International Physical Activity Questionnaires (IPAQ) | 16 months
  Vigorous activity, moderate activity, walking, and time spent sitting.
  There are two forms of output from scoring the IPAQ. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity. Higher activity levels or more MET minutes per week equates to more physical activity.
Change from 4 months to 16 months on the International Physical Activity Questionnaires (IPAQ) | 16 months
  Vigorous activity, moderate activity, walking, and time spent sitting.
  There are two forms of output from scoring the IPAQ. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity. Higher activity levels or more MET minutes per week equates to more physical activity.
Change from baseline to 4 months on the Charlson comorbidity index | 4 months
  Comorbidity status calculated from from electronic medical record diagnoses. 19 possible conditions as identified in Charlson 1987.
  A weighted index of scores takes into account the presence vs absence of a disease and the seriousness of such disease. Conditions Scores range from 0-37 and depend on how many of the 19 possible conditions the person has and the seriousness of those conditions. Lower scores represent fewer or no comorbidities.
Change from baseline to 16 months on the Charlson comorbidity index | 16 months
  Comorbidity status calculated from from electronic medical record diagnoses
Change from 4 months to 16 months on the Charlson comorbidity index | 16 months
  Comorbidity status calculated from from electronic medical record diagnoses
Change from baseline to 4 months on Hemoglobin A1c | 4 months
  Non-fasting Hemoglobin A1c, measured by the Afinion meter (Alere, Inc., Waltham, MA, USA)
Change from baseline to 16 months on Hemoglobin A1c | 16 months
  Non-fasting Hemoglobin A1c, measured by the Afinion meter (Alere, Inc., Waltham, MA, USA) among participants with diabetes.
Change from 4 months to 16 months on Hemoglobin A1c | 16 months
  Non-fasting Hemoglobin A1c, measured by the Afinion meter (Alere, Inc., Waltham, MA, USA) among participants with diabetes.
Change from baseline to 4 months on Lipid profile (Triglycerides, HDL, LDL, Total) | 4 months
  Non-fasting lipid profile measured by Cholestech meter (Alere, Inc.)
Change from baseline to 4 months on systolic/diastolic blood pressure | 4 months
  Seated and resting blood pressure
Change from 4 months to 16 months on systolic/diastolic blood pressure | 16 months
  Seated and resting blood pressure
Change from baseline to 16 months on systolic/diastolic blood pressure | 16 months
  Seated and resting blood pressure
Change from baseline to 4 months on Coronary heart disease risk | 4 months
  Calculated from Framingham risk score LDL points total. Coronary heart disease risk scores are the 10-year congenital heart disease risk. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.
Change from baseline to 16 months on Coronary heart disease risk | 16 months
  Calculated from Framingham risk score LDL points total. Coronary heart disease risk scores are the 10-year congenital heart disease risk. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.
Change from 4 months to 16 months on Coronary heart disease risk | 16 months
  Calculated from Framingham risk score LDL points total. Coronary heart disease risk scores are the 10-year congenital heart disease risk. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.
Change from baseline to 4 months on diabetes risk | 4 months
  Calculated from European prospective investigation into cancer and nutrition (EPIC) diabetes risk score. Diabetes risk scores of 534-585 and 586-657 are associated with 3.0-4.9% and 5.0-9.9% incidence of diabetes within five years, respectively.
Change from baseline to 16 months on diabetes risk | 16 months
  Calculated from European prospective investigation into cancer and nutrition (EPIC) diabetes risk score. Diabetes risk scores of 534-585 and 586-657 are associated with 3.0-4.9% and 5.0-9.9% incidence of diabetes within five years, respectively.
Change from 4 months to 16 months on diabetes risk | 4 months
  Calculated from European prospective investigation into cancer and nutrition (EPIC) diabetes risk score. Diabetes risk scores of 534-585 and 586-657 are associated with 3.0-4.9% and 5.0-9.9% incidence of diabetes within five years, respectively.
Change from baseline to 4 months on dietary intake based on Block 2005 food frequency questionnaire Spanish version | 4 months
  Usual and customary intake of a wide array of nutrients and food groups Dietary intake of sugar (g), sodium (mg), saturated fat (g), vegetables (servings), and fruit (servings) was reported. Generally, higher intake of sugar, sodium, and saturated fat and lower fruit/vegetable intake is associated with poor dietary intake patterns.
Change from 4 months to 16 months on patient activation measured using Patient Activation Measure 13 | 16 months
  One's knowledge of, skills in, and confidence in health self-management.
  PAM 13 scores can theoretically range from 0-100. Higher PAM scores are related to more desirable outcome.
Pain measured using Brief Pain Inventory short form | 16 months
  Pain is comprised of a severity and interference subscore. The severity subscale measures amount of pain a person has experienced at its "worst," "least," and "average" levels, as well as present pain. The interference subscale assesses how much a person's pain interferes with everyday life.
Heart healthy behaviors measured using the My Habits questionnaire | 16 months
  Measure of heart healthy behaviors within 3 subscales: salt intake, fat and cholesterol consumption, and weight control behaviors. A 4-point Likert scale (1=never, 4=always) is used to answer "How often have you done the following over the past month?" Responses are summed and averaged for each subscale; higher scores represent healthier habits.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No plans were made to share data publicly as this was not a government-funded study.

REFERENCES:
- [Background] Schepens Niemiec SL, Blanchard J, Vigen CLP, Martinez J, Guzman L, Concha A, Fluke M, Carlson M. Evaluation of inverted exclamation markVivir Mi Vida! to improve health and wellness of rural-dwelling, late middle-aged Latino adults: results of a feasibility and pilot study of a lifestyle intervention. Prim Health Care Res Dev. 2018 Sep;19(5):448-463. doi: 10.1017/S1463423617000901. Epub 2018 May 6. PMID 29729677
- [Background] Schepens Niemiec SL, Blanchard J, Vigen CLP, Martinez J, Guzman L, Fluke M, Carlson M. A Pilot Study of the inverted exclamation markVivir Mi Vida! Lifestyle Intervention for Rural-Dwelling, Late-Midlife Latinos: Study Design and Protocol. OTJR (Thorofare N J). 2019 Jan;39(1):5-13. doi: 10.1177/1539449218762728. Epub 2018 Mar 7. PMID 29514544
- [Background] Schepens Niemiec SL, Vigen CLP, Martinez J, Blanchard J, Carlson M. Long-Term Follow-Up of a Lifestyle Intervention for Late-Midlife, Rural-Dwelling Latinos in Primary Care. Am J Occup Ther. 2021 Mar-Apr;75(2):7502205020p1-7502205020p11. doi: 10.5014/ajot.2021.042861. PMID 33657344

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT04623489/Prot_SAP_000.pdf